CLINICAL TRIAL: NCT05875701
Title: A Phase 3 Study to Evaluate the Immunogenicity and Safety of Novavax COVID-19 Vaccine(s) as Second or Subsequent Booster After mRNA Vaccines in Individuals 18 to 49 Years of Age
Brief Title: Phase 3 Study of Novavax Vaccine(s) as Booster Dose After mRNA Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019nCoV-312
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NVX CoV2373 (Ancestral strain) (Experimental): 1dose of NVX-COV2373 on Day 1
  Interventions: Biological: NVX-CoV2373
- Updated COVID-19 Vaccine (Experimental): 1dose of updated COVID-19 vaccine on Day 1
  Interventions: Biological: SARS-CoV-2 rS antigen/Matrix-M Adjuvant

INTERVENTIONS:
Biological: NVX-CoV2373 — 1 intramuscular (IM) injection of 5 µg SARS-CoV-2 rS + 50 µg Matrix-M1 adjuvant (0.5 mL) given on Day 1
  Other Names: SARS-CoV-2 rS/Matrix-M Adjuvant
  Arms: NVX CoV2373 (Ancestral strain)
Biological: SARS-CoV-2 rS antigen/Matrix-M Adjuvant — 1 intramuscular (IM) injection of 5 µg SARS-CoV-2 rS antigen+ 50 µg Matrix-M1 adjuvant (0.5 mL) given on Day 1
  Other Names: Updated Novavax COVID-19 vaccine
  Arms: Updated COVID-19 Vaccine

SUMMARY:
This is an open-label Phase 3 study evaluating the immunogenicity and safety of Novavax vaccine(s) with Matrix-M™ adjuvant (ancestral strain NVX-CoV2373 and an alternative strain and/or multivalent Novavax vaccine) as booster doses following a series of primary and booster doses of authorized/approved mRNA vaccines followed by a single booster dose of NVX-CoV2373 in the Novavax 2019nCoV-307 study (NCT05463068).

DETAILED DESCRIPTION:
This Phase 3 study investigates the immunogenicity and safety of Novavax's NVX-CoV2373 vaccine (including its Matrix-M adjuvant) as an additional booster dose for adults aged 18 to 49. Participants must have already received both their primary mRNA vaccine series and at least one booster dose of the same type. All participants were previously enrolled in Study 307 (NCT05463068), where they received either their primary mRNA vaccines with or without an additional mRNA booster, followed by a single NVX-CoV2373 booster.

The study involves up to 300 volunteers who will receive a single dose of the Novavax vaccine (5 micrograms of recombinant spike protein antigen and 50 micrograms of Matrix-M adjuvant) on Day 1.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all the following criteria:

1. Adults 18 to 49 years (inclusive) of age at the time of vaccination in Study 307 who received two or three doses of mRNA prior to enrollment in Study 307, then one dose of ancestral strain NVX-CoV2373 in Study 307.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of study (EOS) visit OR agree to consistently use a medically acceptable method of contraception from at least 28 days prior to enrollment and through the EOS visit.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the study vaccination.
5. Agree to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study. Note: For participants who become hospitalized with COVID-19, participation in investigational treatment studies is permitted.
6. Documented receipt of COVID-19 vaccines. The most recent dose of NVX-CoV2373 must have been administered at least 180 days prior to vaccination in this study.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study.

1. Received any additional COVID-19 vaccine booster after the Day 1 dose of NVX-CoV2373 administered during participation in Study 307.
2. History of laboratory-confirmed (by polymerase chain reaction [PCR] or rapid antigen test) COVID-19 infection ≤ 4 months prior to Day 1.
3. Current participation in research involving receipt of an investigational product (drug/biologic/device).
4. Any known allergies or history of anaphylaxis to the active substance or any of the other ingredients contained in the investigational product.
5. Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) or therapy that causes clinically significant immunosuppression.
6. Received any vaccine ≤ 90 days prior to study vaccination, except for influenza vaccine which may be received > 4 days prior to study vaccine, or rabies vaccine, which may be received at any time if medically indicated.
7. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination, except for rabies immunoglobulin which may be given if medically indicated.
8. Active cancer (malignancy) on chemotherapy that is judged to cause significant immunocompromise within 1 year prior to first study vaccination (with the exception of malignancy cured via excision, at the discretion of the investigator).
9. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the EOS visit.
10. Suspected or known history of alcohol abuse or drug addiction within 3 months prior to the study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
11. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
12. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
13. Participants with a history of myocarditis or pericarditis.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (5):
- United States (5):
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Research Your Health, Plano, Texas
  - Tekton Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- NVX-CoV2540(Updated COVID-19 Vaccine): 1dose of updated COVID-19 vaccine on Day 1
  SARS-CoV-2 rS antigen/Matrix-M Adjuvant: 1 intramuscular (IM) injection of 5 µg SARS-CoV-2 rS antigen+ 50 µg Matrix-M1 adjuvant (0.5 mL) given on Day 1
Period: Overall Study
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Started | 104 | 43
Completed | 101 | 42
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine) | Total
Number analyzed (Participants) | 104 | 43 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (7.97) | 37.2 (9.20) | 37.75 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 23 | 86
  Male | 41 | 20 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 92 | 36 | 128
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 25 | 98
  Black or African American | 23 | 15 | 38
  Asian | 3 | 3 | 6
  Other | 3 | 0 | 3
  Not Reported/Specified | 2 | 0 | 2
Time between first dose of previous NVX vaccine at Study 307 and Day 1 dose of Study 312 [Mean (Standard Deviation); unit: days] | 265.0 (25.92) | 311.0 (1.85) | 288 (27.77)
PCR, n (%) [Count of Participants; unit: Participants]
  Positive | 1 | 0 | 1
  Negative | 98 | 42 | 140
  Missing | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Neutralizing Antibody (Nab) for SARS-CoV-2 Wildtype Virus (Wuhan) Responses Expressed as Geometric Mean Titers (GMT)
Description: Neutralizing Antibody responses to ancestral strain Novavax vaccine (NVX-CoV2373) for the participants in the ancestral strain NVX-2373 group and NVX-CoV2540 group at Day 29
Time Frame: Day 28
Population: Per Protocol Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 98 | 40
titers
  Date of 1st booster dose (Study 307) | 173.2 [123.0 to 243.8] | 159.5 [94.3 to 269.9]
  28 days after 1st booster dose (Study 307) | 396.6 [328.7 to 478.6] | 436.0 [305.6 to 622.2]
  Date of 2nd booster dose (Study 312) | 306.4 [222.6 to 421.6] | 420.7 [282.5 to 626.6]
  28 days after 2nd booster dose (Study 312) | 393.2 [318.0 to 486.2] | 835.0 [597.1 to 1167.6]

2. Secondary Outcome: Neutralizing Antibody (Nab) for SARS-CoV-2 Wildtype Virus (Wuhan) Responses Expressed as Seroconversion Rate (SCR)
Description: Neutralizing Antibody responses to ancestral strain Novavax vaccine (NVX-CoV2373) for the participants in the ancestral strain NVX-2373 group and NVX-CoV2540 group at Day 28
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 98 | 40
participants
  28 days after 1st booster relative to date of 1st booster | 24 | 11
  28 days after 2nd booster relative to date of 2nd booster | 21 | 11
  28 days after 2nd booster relative to date of 1st booster | 31 | 22

3. Secondary Outcome: Serum Immunoglobulin G (IgG) ELISA Units to SARS-CoV-2 Spike Protein (Wuhan) Expressed as Geometric Mean ELISA Unit (GMEU)
Description: Serum Immunoglobulin G (IgG) ELISA Units to SARS-CoV-2 Spike Protein (Wuhan) in Ancestral strain NVX-CoV2373 group and updated NVX Vaccine group at Day 28
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: Elisa Units per mL
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 98 | 40
Elisa Units per mL
  Date of 1st booster dose (Study 307) | 37822.4 [29104.7 to 49151.4] | 32446.8 [22453.4 to 46888.0]
  28 days after 1st booster dose (Study 307) | 93969.2 [79844.0 to 110593.4] | 93636.6 [69077.5 to 126927.1]
  Date of 2nd booster dose (Study 312) | 67333.6 [54380.8 to 83371.6] | 71336.1 [50460.2 to 100848.6]
  28 days after 2nd booster dose (Study 312) | 162144.7 [136476.6 to 192640.4] | 203864.0 [148535.6 to 279801.8]

4. Secondary Outcome: Serum Immunoglobulin G (IgG) ELISA Units to SARS-CoV-2 Spike Protein (Wuhan) Expressed as SCR
Description: as for outcome 3
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 98 | 40
participants
  28 days after 1st booster relative to date of 1st booster | 22 | 11
  28 days after 2nd booster relative to date of 2nd booster | 22 | 11
  28 days after 2nd booster relative to date of 1st booster | 45 | 22

5. Secondary Outcome: Neutralizing Antibody Responses (Post-Booster) Expressed as GMT
Description: Post Booster Neutralizing Antibody responses GMTs compared with post-first booster results from Study 307
Time Frame: Day 0 and Day 28 of Study 307 and Study 312 (approximately 1 year from Day 0 of Study 307 and Day 0 of Study 312)
Population: Study 307 results represent results from a prior study in which participants took part in.
  Study 312 refers to the study in this specific record.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- NVX CoV2373 (Ancestral Strain): NVX-CoV2373: 1 intramuscular (IM) injection of 5 µg SARS-CoV-2 rS + 50 µg Matrix-M1 adjuvant (0.5 mL)
Arm/Group | NVX CoV2373 (Ancestral Strain)
Number analyzed (Participants) | 98
geometric mean titer
  Day 0 of 1st booster dose (Study 307) | 173.2 [123.0 to 243.8]
  28 days after 1st booster dose (Study 307) | 396.6 [328.7 to 478.6]
  Day 0 of 2nd booster dose (Study 312) | 306.4 [222.6 to 421.6]
  28 days after 2nd booster dose (Study 312) | 393.2 [318.0 to 486.2]

6. Secondary Outcome: Serum IgG Antibody Levels (Post-Booster) Expressed as GMEU
Description: Post Booster Serum IgG antibody levels expressed GMEUs compared with post-first booster results from Study 307
Time Frame: Day 0 and Day 28 of Study 307 and Study 312 (approximately 1 year from Day 0 of Study 307 and Day 0 of Study 312)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean Elisa Units
Arm/Group | NVX CoV2373 (Ancestral Strain)
Number analyzed (Participants) | 98
geometric mean Elisa Units
  Day 0 of 1st booster dose (Study 307) | 37822.4 [29104.7 to 49151.4]
  28 days after 1st booster dose (Study 307) | 93969.2 [79844.0 to 110593.4]
  Day 0 of 2nd booster dose (Study 312) | 67333.6 [54380.8 to 83371.6]
  28 days after 2nd booster dose (Study 312) | 162144.7 [136476.6 to 192640.4]

7. Secondary Outcome: Human Angiotensin-Converting Enzyme 2 (hACE2) Receptor Binding Inhibition Assay Expressed as SCR
Description: hACE2 Receptor Binding Inhibition Assay the SARS-CoV-2 ancestral strain spike protein expressed as SCR at Day 28
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NVX CoV2373 (Ancestral Strain)
Number analyzed (Participants) | 98
Percentage of participants | 12.6 [5.9 to 21.2]

8. Secondary Outcome: Number of Participants Reported Solicited Local and Systemic Adverse Events (AEs)
Description: Number of participants reported Solicited Local and Systemic Adverse Events (AEs) in the 7 days following study vaccination.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 104 | 43
Participants
  Any solicited local reaction | 68 | 31
  Pain | 48 | 18
  Tenderness | 62 | 29
  Redness | 7 | 1
  Swelling | 5 | 0
  Systemic reaction | 69 | 24
  Fever | 1 | 1
  Fatigue | 49 | 11
  Malaise | 31 | 5
  Muscle pain | 43 | 19
  Joint pain | 19 | 7
  Nausea/vomiting | 12 | 5
  Headache | 40 | 13

9. Secondary Outcome: Number of Participants Reported With Medically Attended Adverse Events (MAAEs)
Description: Number of participants reported with Medically Attended Adverse Events (MAAEs) through Day 180 after the vaccine dose.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 104 | 43
Participants
  MAAEs | 5 | 1
  Severe MAAEs | 0 | 1

10. Secondary Outcome: Number of Participants Reported With Serious Adverse Events (SAEs)
Description: Number of participants reported with Serious Adverse Events (SAEs) through Day 180 after the vaccine dose
Time Frame: Day 1 to Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 104 | 43
Participants | 0 | 1

11. Secondary Outcome: Neutralizing Antibody Responses (Post-Booster) Expressed as GMT
Description: Post Booster Neutralizing Antibody responses GMTs compared with post-first booster results from Study 307
Time Frame: Day 0 and Day 28 of Study 307 and Study 312 (approximately 1 year from Day 0 of Study 307 and Day 0 of Study 312)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 40
geometric mean titer
  Day 0 of 1st booster dose (Study 307) | 159.5 [94.3 to 269.9]
  28 days after 1st booster dose (Study 307) | 436.0 [305.6 to 622.2]
  Day 0 of 2nd booster dose (Study 312) | 420.7 [282.5 to 626.6]
  28 days after 2nd booster dose (Study 312) | 835.0 [597.1 to 1167.6]

12. Secondary Outcome: Serum IgG Antibody Levels (Post-Booster) Expressed as GMEU
Description: Post Booster Serum IgG antibody levels expressed GMEUs compared with post-first booster results from Study 307
Time Frame: Day 0 and Day 28 of Study 307 and Study 312 (approximately 1 year from Day 0 of Study 307 and Day 0 of Study 312)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean Elisa Units
Arm/Group | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 40
geometric mean Elisa Units
  Day 0 of 1st booster dose (Study 307) | 32446.8 [22453.4 to 46888.0]
  28 days after 1st booster dose (Study 307) | 93636.6 [69077.5 to 126927.1]
  Day 0 of 2nd booster dose (Study 312) | 71336.1 [50460.2 to 100848.6]
  28 days after 2nd booster dose (Study 312) | 203864.0 [148535.6 to 279801.8]

13. Secondary Outcome: Human Angiotensin-Converting Enzyme 2 (hACE2) Receptor Binding Inhibition Assay Expressed as SCR
Description: hACE2 Receptor Binding Inhibition Assay to the NVX-CoV2540(Updated COVID-19 Vaccine) expressed as SCR at Day 28
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | NVX-CoV2540(Updated COVID-19 Vaccine)
Number analyzed (Participants) | 40
participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | NVX CoV2373 (Ancestral Strain) | NVX-CoV2540(Updated COVID-19 Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/104 | 1/43
Other Adverse Events (participants affected / at risk) | 2/104 | 1/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVX CoV2373 (Ancestral Strain) (N=104) | NVX-CoV2540(Updated COVID-19 Vaccine) (N=43)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVX CoV2373 (Ancestral Strain) (N=104) | NVX-CoV2540(Updated COVID-19 Vaccine) (N=43)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT05875701/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05875701/SAP_001.pdf